CLINICAL TRIAL: NCT01486134
Title: Pilot Study of Real Time MR Temperature Monitoring of Multipolar Radiofrequency Ablation of Large Hepatocellular Carcinomas (≥ 5 CM)-ARMTICH STUDY
Brief Title: Major RF Ablations of Hepatomas Under MR Thermometry Monitoring
Acronym: ARMTICH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For technical reasons
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100138/AOM 10266; 2011-A00007-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2011-11-22; First posted 2011-12-06 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Cancer
Keywords: Hepatocellular carcinoma; Radiofrequency ablation; Multipolar mode; Recurrence; Cirrhosis; MR temperature monitoring; large tumor
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Recurrence; Fibrosis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- procedure (Experimental)
  Interventions: Procedure: Multipolar Radiofrequency ablation

INTERVENTIONS:
Procedure: Multipolar Radiofrequency ablation — Percutaneous multipolar radiofrequency ablation.
  Other Names: Radiofrequency ablation

SUMMARY:
Object of the study:

To assess the effectiveness of MR temperature monitoring of RFA of large hepatocellular carcinomas (HCC) (≥ 5 cm) in terms of complete tumor necrosis rate achieved and in term of reduction of the number of procedure required to obtain complete ablation of the tumors.

Experimental plan :

This pilot study consist to perform in a single center a single procedure of the multipolar RF ablation under MR temperature monitoring for the treatment of up to three HCC with diameter ranging from 5 cm and 10 cm in 20 inoperable patients. The main judgement criterion of the study will be the rate of complete ablation one month after one RFA procedure performed under MR temperature monitoring. The secondary criteria are, the 2-years local recurrence rate (after the first initial RF ablation procedure performed under MR temperature imaging ± additional RF ablation procedures under ultrasound monitoring in case of remnant viable foci of tumor), the potential reduction of the number of RF procedures required to achieve complete necrosis and the complication rate of RF ablation procedure performed under MR temperature monitoring.

In exploratory attempt, the study will include comparative assessment of these criteria with a historic leg of patients previously treated by the same operator in the same center for similar large tumor by multipolar RFA but using exclusively ultrasound monitoring.

DETAILED DESCRIPTION:
The RF procedure and results assessment:

1. In preparing MR room, the patient will be positioned on MR bed put on dedicated MR compatible trolley. The abdominal antenna will be installed.
2. General anesthesia with tracheal intubation will be performed.
3. Up to six RF electrodes (up to 6 depending on the size and the location of the tumor) will be inserted under ultrasound guidance.
4. The patient will be translated without any direct manipulation in the magnet.
5. With usual T1 and T2 weighted MR morphologic sequences the poisoning of electrode will be checked and if necessary adjusted
6. Adjustment or MR temperature imaging (before RF energy deposition)
7. Starting of RF procedure under MR temperature monitoring
8. According to thermal dose maps data repositioning of electrodes and complementary energy deposition if necessary
9. Hot withdrawal of electrodes
10. Immediate (T0) post procedure MR assessment of the limits of ablation zone (T2 SPIRCHOL, Diffusion B600, In out phase, THRIVE dynamic after intravenous gadolinium injection).

After the procedure patients will be monitored at least 48 h.

MR assessment of treatment response will be performed one month after the procedure (same MR protocol performed at T0).

If the ablation is complete follow up will be ensured by MR every three months. If the ablation appeared incomplete or in case of recurrence additional RF ablation will be performed if the patient stills met the criteria of the treatment. The eventual additional RF ablation will be performed under ultrasound monitoring (the response to each additional RF ablation procedure will be assessed by MR one month after).

At the end of the study patients for whom complete radiological response of the tumor(s) initially treated (not local or distance recurrences) will be never achieved, will be considered in treatment failure.

Local recurrence is defined as the reappearance of viable tumor in contact of ablation zone of a tumor considered at least on one MR post therapeutic examination as completely ablated.

All the adverse effect and complication will be recorded and reported.

Quantitative analysis of 2D and 3D parameters of tumors and their related ablation zones as observed at the end of RF procedures on temperature maps using thermal dose concept (as previously extensively investigated) and with usual morphologic MR imaging (all used sequences) before, during and after the procedure (one month after) will be recorded and compared.

Antibioprophylaxy: will be prescribed in patients with an antecedent of endoscopic sphincterotomy (according to the CLIN protocol of Jean Verdier Hospital) and will be extended in patients : 1 older than 75 years , 2 patient with vesicular lithiasis 3) patients with nodule previously treated by embolization and those with a severe diabetes

ELIGIBILITY:
Inclusion Criteria:

* Patient of 18 year old.
* Up to 3 tumors unresectable suspected to be HCC according the criteria as previously defined by EASL and recently revised by AASLD among them at least one having a maximal diameter equal or larger than 5 cm.
* Proof of underlying cirrhosis.
* Multidisciplinary decision of RF ablation treatment
* Informed consent of patient
* Available healthcare insurance

Exclusion Criteria:

* Patient with short term life training uncontrollable disease
* Pregnancy
* Follow up Impossible
* Contra indication for general anesthesia
* Contra indication for MR examination with gadolinium injection
* Tumor located at less than 10 mm from colonic wall or main biliary tract
* Tumor invisible on MR examination
* Absence of safe percutaneous course to puncture the tumor
* Child - Pugh B or C cirrhosis
* Abundant ascites
* PROTHROMBIN activity < 50 %
* Platelet count < 40 .10 3/ml
* Antecedent of ascitis decompensation
* Severe portal hypertension defined by the presence of large oesophageal variceal (grade 2) , of radiological ascitis or umbilical vein repermeabilisation
* Elevation of transaminases (>3 upper limit normal range)
* Antecedent of biliodigestive anastomosis
* Antecedent of endoscopic sphincterotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Rate of complete ablation one month after one RFA procedure | One month after one RFA procedure

SECONDARY OUTCOMES:
2-years local recurrence rate | 2 years
Number of procedure required to achieve complete ablation | One month after completion of treatment course
Primary treatment effectiveness (assessed 1 month after completion of treatment course which can include up to 3 RFA procedures performed monthly) | 1 month after completion of treatment
Complication rate per RF procedure under MR temperature monitoring | 2 years
Agreement of 2D and 3D measurements of ablations zones on IRMT° images and those measured on conventional magnitude MR images. | during and after the procedure (one month after)

CONTACTS AND LOCATIONS:
Overall Officials: SEROR Olivier, MD-PHD, Principal Investigator — CHU Jean VERDIER-Radiology department
Locations (1):
- CHU Jean VERDIER, Bondy, France

REFERENCES:
- [Background] N'Kontchou G, Mahamoudi A, Aout M, Ganne-Carrie N, Grando V, Coderc E, Vicaut E, Trinchet JC, Sellier N, Beaugrand M, Seror O. Radiofrequency ablation of hepatocellular carcinoma: long-term results and prognostic factors in 235 Western patients with cirrhosis. Hepatology. 2009 Nov;50(5):1475-83. doi: 10.1002/hep.23181. PMID 19731239
- [Background] Seror O, N'Kontchou G, Ibraheem M, Ajavon Y, Barrucand C, Ganne N, Coderc E, Trinchet JC, Beaugrand M, Sellier N. Large (>or=5.0-cm) HCCs: multipolar RF ablation with three internally cooled bipolar electrodes--initial experience in 26 patients. Radiology. 2008 Jul;248(1):288-96. doi: 10.1148/radiol.2481071101. Epub 2008 May 15. PMID 18483229
- [Background] Seror O, Lepetit-Coiffe M, Quesson B, Trillaud H, Moonen CT. Quantitative magnetic resonance temperature mapping for real-time monitoring of radiofrequency ablation of the liver: an ex vivo study. Eur Radiol. 2006 Oct;16(10):2265-74. doi: 10.1007/s00330-006-0210-9. Epub 2006 Apr 11. PMID 16607496
- [Background] Seror O, Lepetit-Coiffe M, Le Bail B, de Senneville BD, Trillaud H, Moonen C, Quesson B. Real time monitoring of radiofrequency ablation based on MR thermometry and thermal dose in the pig liver in vivo. Eur Radiol. 2008 Feb;18(2):408-16. doi: 10.1007/s00330-007-0761-4. Epub 2007 Sep 26. PMID 17899103
- [Background] Lepetit-Coiffe M, Laumonier H, Seror O, Quesson B, Sesay MB, Moonen CT, Grenier N, Trillaud H. Real-time monitoring of radiofrequency ablation of liver tumors using thermal-dose calculation by MR temperature imaging: initial results in nine patients, including follow-up. Eur Radiol. 2010 Jan;20(1):193-201. doi: 10.1007/s00330-009-1532-1. Epub 2009 Aug 6. PMID 19657650